CLINICAL TRIAL: NCT02092220
Title: A Multicenter Study of Outpatient Automated Blood Glucose Control With a Bihormonal Bionic Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Multicenter Study
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Bionic Pancreas; Insulin; Glucagon; Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bionic Pancreas (Experimental): Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin and glucagon using a continuous glucose monitoring (CGM) device, for 11 days.
  Interventions: Device: Bionic Pancreas
- Usual Care (Active Comparator): Usual Care diabetes management, standard of care for diabetes including use of an insulin pump with or without CGM according to the participant's usual practice, for 11 days.
  Interventions: Device: Insulin pump with or without CGM

INTERVENTIONS:
Device: Bionic Pancreas
  Arms: Bionic Pancreas
Device: Insulin pump with or without CGM
  Arms: Usual Care

SUMMARY:
This study will test the hypothesis that a wearable bionic pancreas system that automatically delivers insulin and glucagon can provide superior regulation of glycemia versus usual care for adults with type 1 diabetes.

Please note that all participants must work or attend school at one of the following campuses: Massachusetts General Hospital in Boston, MA; University of Massachusetts Medical Center in Worcester, MA; University of North Carolina in Chapel Hill, NC; Stanford University in Palo Alto, CA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and have had clinical type 1 diabetes for at least one year
* Diabetes managed using an insulin pump for ≥ 6 months
* Prescription medication regimen stable for > 1 month (except for medications that will not affect the safety of the study and are not expected to affect any outcome of the study, in the judgement of the site principal investigator).
* Employee or student working or studying during most of the week at one of the participating campuses (Massachusetts General Hospital in Boston, MA; University of Massachusetts Medical Center in Worcester, MA; University of North Carolina in Chapel Hill, NC; Stanford University in Palo Alto, CA)
* Lives within a 30 minute drive-time radius of the central monitoring location for one of the study sites
* Willing to remain within a 60 minute drive-time radius of the central monitoring location for one of the study sites during each of the 11-day study arms
* Have someone over 18 years of age who lives with them, has access to where they sleep, is willing to be in the house when the subject is sleeping, and is willing to receive calls from the study staff and check the welfare of the study subject if telemetry shows a technical problem or severe biochemical hypoglycemia without subject response and the subject does not answer their telephone (up to two individuals can share this role, but they must be willing to carefully coordinate with each other and the subject so that one of them is clearly designated as having this responsibility at any given time)
* Willing to wear two infusion sets and continuous glucose monitor (CGM) sensor and change sets frequently (at least one new glucagon infusion set daily)

Exclusion Criteria:

* Unable to provide informed consent (e.g. impaired cognition or judgment)
* Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory, unable to speak and read English)
* Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the subject
* Pregnancy [positive urine human chorionic gonadotropin (HCG)] breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception
* Need to go outside of the designated geographic boundaries during either arm of the study
* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days), use of marijuana within 1 month of enrollment, or other substance abuse (use within the last 6 months of controlled substances other than marijuana without a prescription)
* Unwilling or unable to refrain from drinking more than 2 drinks in an hour or more than 4 drinks in a day or use of marijuana during the trial
* Unwilling or unable or to avoid use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of beta blockers will be allowed as long as the dose is stable and the subject does not meet the criteria for hypoglycemia unawareness while taking that stable dose, but use of benzodiazepines or narcotics, even if by prescription, may be excluded according to the judgment of the principal investigator)
* History of liver disease that is expected to interfere with the anti-hypoglycemia action of glucagon (e.g. liver failure or cirrhosis). Other liver disease (i.e. active hepatitis, steatosis, active biliary disease, any tumor of the liver, hemochromatosis, glycogen storage disease) may exclude the subject if it causes significant compromise to liver function or may do so in an unpredictable fashion.
* Renal failure on dialysis
* Personal history of cystic fibrosis, pancreatitis, pancreatic tumor, or any other pancreatic disease besides type 1 diabetes
* Any known history of coronary artery disease including, but not limited to, history of myocardial infarction, stress test showing ischemia, history of angina, or history of intervention such as coronary artery bypass grafting, percutaneous coronary intervention, or enzymatic lysis of a presumed coronary occlusion)
* Abnormal electrocardiogram (EKG) consistent with coronary artery disease or increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, prior myocardial infarction, proximal left anterior descending coronary artery (LAD) critical stenosis (Wellen's sign), prolonged QT interval (> 440 ms). Non-specific ST segment and T wave changes are not grounds for exclusion in the absence of symptoms or history of heart disease. A reassuring evaluation by a cardiologist after an abnormal EKG finding may allow participation.
* Congestive heart failure (CHF) [established history of CHF, lower extremity edema, paroxysmal nocturnal dyspnea, or orthopnea]
* History of transient ischaemic attack (TIA) or stroke
* Seizure disorder, history of any non-hypoglycemic seizure within the last two years, or ongoing treatment with anticonvulsants
* History of hypoglycemic seizures or coma in the last year
* History of pheochromocytoma: fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor:

  * episodic or treatment refractory (requiring 4 or more medications to achieve normotension) hypertension
  * paroxysms of tachycardia, pallor, or headache
  * personal or family history of multiple endocrine neoplasia type 2A (MEN 2A), multiple endocrine neoplasia type 2B (MEN 2B), neurofibromatosis, or von Hippel-Lindau disease
* History of adrenal disease or tumor
* Hypertension with systolic blood pressure (BP) ≥160 mm Hg or diastolic BP ≥100 despite treatment
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to radio-frequency (RF) interference
* Unable to completely avoid acetaminophen for duration of study
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study
* History of eating disorder such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
* History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
* Use oral [e.g. thiazolidinediones, biguanides, sulfonylureas, glitinides, dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium-glucose co-transporter 2 (SGLT-2) inhibitors] anti-diabetic medications
* Lives in or frequents areas with poor Verizon wireless network coverage (which would prevent remote monitoring)
* Any factors that, in the opinion of the site principal investigator or overall principal investigator, would interfere with the safe completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Massachusetts General Hospital (MGH) Diabetes Research Center, Boston, Massachusetts
  - UMass Medical Center, Worcester, Massachusetts
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Result] El-Khatib FH, Balliro C, Hillard MA, Magyar KL, Ekhlaspour L, Sinha M, Mondesir D, Esmaeili A, Hartigan C, Thompson MJ, Malkani S, Lock JP, Harlan DM, Clinton P, Frank E, Wilson DM, DeSalvo D, Norlander L, Ly T, Buckingham BA, Diner J, Dezube M, Young LA, Goley A, Kirkman MS, Buse JB, Zheng H, Selagamsetty RR, Damiano ER, Russell SJ. Home use of a bihormonal bionic pancreas versus insulin pump therapy in adults with type 1 diabetes: a multicentre randomised crossover trial. Lancet. 2017 Jan 28;389(10067):369-380. doi: 10.1016/S0140-6736(16)32567-3. Epub 2016 Dec 20. PMID 28007348

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 participants were enrolled in the trial, but only 43 participants actually participated. 2 participants were not eligible and 3 participants were not randomized because target enrollment was already met.
Groups:
- Bionic Pancreas Then Usual Care: Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin and glucagon using a continuous glucose monitoring (CGM) device, for 11 days in Period 1 followed by Usual Care diabetes management, standard of care for diabetes including use of an insulin pump with or without CGM according to the participant's usual practice, for 11 days in Period 2. There was a 3 to 10-day washout period between periods.
- Usual Care Then Bionic Pancreas: Usual Care diabetes management, standard of care for diabetes including use of an insulin pump with or without CGM according to the participant's usual practice, for 11 days in Period 1 followed by Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin and glucagon using a continuous glucose monitoring (CGM) device, for 11 days in Period 2. There was a 3 to 10-day washout period between periods.
Period: Period 1
Arm/Group | Bionic Pancreas Then Usual Care | Usual Care Then Bionic Pancreas
Started | 21 | 22
Completed | 21 | 20
Not Completed | 0 | 2
Not completed — Unrelated Illness | 0 | 2
Period: Period 2
Arm/Group | Bionic Pancreas Then Usual Care | Usual Care Then Bionic Pancreas
Started | 21 | 20
Completed | 20 | 19
Not Completed | 1 | 1
Not completed — Severe Hypoglycaemia | 1 | 0
Not completed — Nausea, Anxiety, Inconvenience | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants who completed both periods of the study.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Continuous Glucose Monitoring Glucose (CGMG) Values During Days 2 to 11
Description: Glucose reading were taken every 5 minutes by the CGM. The glucose results on Days 2 to 11 were averaged.
Time Frame: Days 2 to 11 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
milligrams/deciliter (mg/dL) | 141.2 (9.9) | 161.5 (28.7)
Statistical Analysis 1: Comparison: Bionic Pancreas vs Usual Care; Test type: Superiority; p < 0.0001, t-test, 2 sided — Repeated measures model; Mean Difference (Final Values) = -20.28, 95% CI 2-sided [-28.00 to -12.56], Standard Deviation 24.59 — Bionic Pancreas Arm - Usual Care Arm

2. Primary Outcome: Percentage of Time Spent With CGMG Concentration < 60 mg/dL During Days 2 to 11
Description: Glucose reading were taken every 5 minutes by the CGM.The percentage of time that the glucose concentration was less than 60 mg/dL [3.3 millimoles/liter (mmol/L)] during Days 2 to 11 was calculated.
Time Frame: Days 2 to 11 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
percentage of time | 0.6 (0.6) | 1.9 (1.7)
Statistical Analysis 1: Comparison: Bionic Pancreas vs Usual Care; Test type: Superiority; p < 0.0001, t-test, 2 sided — Repeated measures model; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.8 to 1.8]

3. Secondary Outcome: Mean CGMG Values
Description: Glucose reading were taken every 5 minutes by the CGM. The glucose results on Days 1 and Days 1 to 11 were averaged.
Time Frame: Day 1 and Days 1 to 11 in each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
mg/dL
  Day 1 | 145.3 (17.6) | 161.9 (45.2)
  Days 1 to 11 | 141.5 (10.0) | 161.7 (29.3)

4. Secondary Outcome: Percentage of Time With CGMG Concentration by Ranges During Day 1
Description: Glucose reading were taken every 5 minutes by the CGM.The percentage of time that the glucose concentration was less than the following ranges were calculated:
  < 50 mg/dL (2.8 mmol/L) < 60 mg/dL (3.3 mmol/L) < 70 mg/dL (3.9 mmol/L) 70 to 120 mg/dL (3.9 to 6.7 mmol/L) 70 to180 mg/dl (3.9 to 10.0 mmol/L) > 180 mg/dL (10.0 mmol/L) > 250 mg/dL (13.9 mmol/L)
Time Frame: Day 1 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
percentage of time
  < 50 mg/dl (2.8 mmol/L) | 0.1 (0.3) | 0.9 (1.5)
  < 60 mg/dL (3.3 mmol/L) | 0.5 (0.9) | 2.3 (3.4)
  < 70 mg/dl (3.9 mmol/L) | 1.5 (2.3) | 5.0 (6.5)
  70 to 120 mg/dL (3.9 to 6.7 mmol/L) | 39.4 (13.6) | 28.5 (18.6)
  70-180 mg/dl (3.9 to 10.0 mmol/L) | 76.8 (11.5) | 62.1 (22.2)
  > 180 mg/dL (10.0 mmol/L) | 21.7 (11.2) | 32.9 (24.0)
  > 250 mg/dL (13.9 mmol/L) | 6.0 (7.4) | 12.3 (17.7)

5. Secondary Outcome: Percentage of Time With CGMG Concentration by Ranges During Days 1 to 11
Description: Glucose reading were taken every 5 minutes by the CGM.The percentage of time that the glucose concentration was less than the following ranges were calculated:
  < 50 mg/dL (2.8 mmol/L) < 70 mg/dL (3.9 mmol/L) 70 to 120 mg/dL (3.9 to 6.7 mmol/L) 70 to180 mg/dl (3.9 to 10.0 mmol/L) > 180 mg/dL (10.0 mmol/L) > 250 mg/dL (13.9 mmol/L)
Time Frame: Days 1 to 11 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
percentage of time
  < 50 mg/dl (2.8 mmol/L) | 0.1 (0.1) | 0.6 (0.6)
  < 60 mg/dL (3.3 mmol/L) | 0.6 (0.5) | 1.9 (1.8)
  < 70 mg/dl (3.9 mmol/L) | 1.8 (1.4) | 4.6 (3.9)
  70 to 120 mg/dL (3.9 to 6.7 mmol/L) | 40.6 (8.0) | 27.5 (11.3)
  70-180 mg/dl (3.9 to 10.0 mmol/L) | 78.3 (6.0) | 61.9 (14.5)
  > 180 mg/dL (10.0 mmol/L) | 19.9 (6.0) | 33.5 (16.5)
  > 250 mg/dL (13.9 mmol/L) | 4.4 (2.7) | 11.0 (10.3)

6. Secondary Outcome: Percentage of Time With CGMG Concentration by Ranges During Days 2 to 11
Description: as for outcome 5
Time Frame: Days 2 to 11 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
percentage of time
  < 50 mg/dl (2.8 mmol/L) | 0.1 (0.2) | 0.6 (0.6)
  < 70 mg/dl (3.9 mmol/L) | 1.8 (1.4) | 4.5 (3.8)
  70 to 120 mg/dL (3.9 to 6.7 mmol/L) | 40.7 (7.8) | 27.4 (11.4)
  70-180 mg/dl (3.9 to 10.0 mmol/L) | 78.4 (6.0) | 61.9 (14.4)
  > 180 mg/dL (10.0 mmol/L) | 19.8 (6.1) | 33.6 (16.4)
  > 250 mg/dL (13.9 mmol/L) | 4.2 (2.7) | 10.9 (10.0)

7. Secondary Outcome: Percentage of Participants With Mean CGMG < 154 mg/dl
Description: Glucose reading were taken every 5 minutes by the CGM. The glucose readings were averaged. 154 mg/dL was the estimated average glucose corresponding to a Glycosylated Hemoglobin A1C of 7%.
Time Frame: Day 1, Days 2 to11, Days 1 to11 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
percentage of participants
  Day 1 | 79 | 59
  Days 1 to 11 | 92 | 41
  Days 2 to 11 | 92 | 41

8. Secondary Outcome: Number of Hypoglycemic Events (< 70 mg/dL, < 60 mg/dL, <50 mg/dL)
Description: A series of hypoglycemic measurements is defined as a single event until there is a break of ≥ 30 minutes between measurements below the defined thresholds of < 70, < 60, and <50 mg/dL.
Time Frame: Days 1-11
Measure: Mean (Standard Deviation); unit: hypoglycemic events
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
hypoglycemic events
  <50 mg/dl | 0.58 (0.87) | 1.0 (1.06)
  <60 mg/dl | 1.33 (1.31) | 2.88 (2.67)
  <70 mg/dl | 2.68 (2.4) | 5.28 (4.14)

9. Secondary Outcome: Percentage of Days That CGM Was Used by Participants as Part of Their Usual Care
Description: The percentage of days that participants reported the CGM device was being worn and working properly is reported.
Time Frame: Days 1-11 of each period
Population: All randomized participants who completed both periods of the study. This outcome measure applies only to the Usual Care arm.
Measure: Number; unit: percentage of days
Arm/Group | Usual Care
Number analyzed (Participants) | 39
percentage of days | 49

10. Secondary Outcome: Glycated Albumin on Day 12
Time Frame: Day 12 of each period
Population: No data was collected for Glycated Albumin.
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: 1,5-anhydroglucitol on Day 12
Time Frame: Day 12 of each period
Population: No data was collected for 1,5-anhydroglucitol.
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Anti-Insulin and Anti-Glucagon Antibodies on Day 12
Time Frame: Day 12 of each period
Population: No data was collected for Anti-Insulin and Anti-Glucagon Antibodies.
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With Severe Hypoglycemic Events
Description: A severe hypoglycemic event is an event where the participant is unable to self-treat and requires the assistance of another person.
Time Frame: 11 days of each period
Population: All participants who completed both periods of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
Participants | 0 | 1

14. Secondary Outcome: Number of Episodes of Symptomatic Hypoglycemia
Description: The number of episodes of symptomatic hypoglycemia were reported daily by the participant. The average number of episodes of symptomatic hypoglycemia per day was calculated.
Time Frame: Day 1, Days 1 to 11 and Days 2 to 11 of each period
Population: All participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: episodes per day
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
episodes per day
  Day 1 | 0.74 (1.04) | 1.13 (1.12)
  Days 1 to 11 | 0.59 (0.56) | 0.90 (0.64)
  Days 2 to 11 | 0.57 (0.54) | 0.88 (0.64)

15. Secondary Outcome: Number of Reported Carbohydrate Interventions for Hypoglycemia
Description: The number of carbohydrate interventions for hypoglycemia were reported daily by the participant. The average number of carbohydrate interventions per day is reported.
Time Frame: Day 1, Days 1 to 11 and Days 2 to 11 of each period
Population: All participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: interventions per day
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
interventions per day
  Day 1 | 0.36 (0.63) | 1.29 (1.25)
  Days 1 to 11 | 0.39 (0.34) | 0.96 (0.72)
  Days 2 to 11 | 0.40 (0.34) | 0.93 (0.72)

16. Secondary Outcome: Total Grams of Carbohydrate Taken for Hypoglycemia
Description: The total grams of carbohydrate taken for hypoglycemia as reported daily by the participant were averaged.
  The total number of grams of carbohydrate taken for hypoglycemia were reported daily by the participant. The total number of grams of carbohydrate taken are reported.
Time Frame: Day 1, Days 1 to 11 and Days 2 to 11 of each period
Population: All participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: grams of carbohydrate per day
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
grams of carbohydrate per day
  Day 1 | 6.18 (11.61) | 25.61 (26.12)
  Days 1 to 11 | 22.04 (13.62) | 34.8 (16.21)
  Days 2 to 11 | 22.27 (13.79) | 34.8 (16.84)

17. Secondary Outcome: Insulin Total Daily Dose
Description: Insulin total daily dose is reported in units per kilogram per day (U/kg/day).
Time Frame: Day 1, Days 1 to 11, Days 2 to 11 of each period
Population: All participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
U/kg/day
  Day 1 | 0.64 (0.20) | 0.64 (0.21)
  Days 1 to 11 | 0.66 (0.15) | 0.63 (0.18)
  Days 2 to 11 | 0.66 (0.15) | 0.62 (0.18)

18. Secondary Outcome: Glucagon Total Daily Dose Levels in the Bionic Pancreas Arm
Description: Glucagon dose level is reported in micrograms per kilogram of body mass per day (µg/kg/day).
Time Frame: Day 1, Days 2 to 11, Days 1 to 11 of each period
Population: All participants who completed both periods of the study. Results are reported for the Bionic Pancreas period only.
Measure: Mean (Standard Deviation); unit: µg/kg/day
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 39
µg/kg/day
  Day 1 | 7.8 (3.84)
  Days 1 to 11 | 6.9 (2.34)
  Days 2 to 11 | 6.8 (2.4)

19. Secondary Outcome: Mean Glucose Target Set by User (Time-weighted Average Over Study Period) in the Bionic Pancreas Arm
Time Frame: Day 1, Days 2 to 11, Days 1 to11, Overall, Daytime, Nighttime of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Bionic Pancreas: All randomized participants who completed both periods of the study.
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 39
mg/dL
  Day 1, Overall | 101.2 (2.0)
  Day 1, Daytime | 101.3 (1.6)
  Day 1, Nighttime | 101.0 (3.9)
  Day 2 to 11, Overall | 101.9 (5.0)
  Day 2 to 11, Daytime | 102.0 (5.1)
  Day 2 to 11, Nighttime | 101.7 (4.9)
  Day 1 to 11, Overall | 101.8 (4.6)
  Day 1 to 11, Daytime | 101.9 (4.7)
  Day 1 to 11, Nighttime | 101.6 (4.5)

20. Secondary Outcome: Percentage of Time Bionic Pancreas Off-line or Not Functioning Properly
Description: Not functioning properly includes issues due to system crash, communication problems between CGM and bionic pancreas, communication problems between bionic pancreas and pumps and pump malfunction.
Time Frame: 11 days
Population: All randomized participants who completed both periods of the study. Reported for the Bionic pancreas arm only
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 39
percentage of time
  Insulin pump Lost Wireless Connectivity | 3.9 (2.5)
  Glucagon Pump Lost Wireless Connectivity | 4.1 (2.4)
  CGM Signal Unavailable | 3.4 (1.3)

21. Secondary Outcome: Mean Nausea Index Score Using a Visual Analog Scale (VAS)
Description: Participants rated their nausea using a 0 to 10 centimeter (cm) VAS where 0=least severe nausea to 10=most severe nausea. The average nausea index scores during Days 1 to 11 and Days 2 to 11 were calculated.
Time Frame: Day 1, Days 1 to 11, Days 2 to 11 and each individual day 2 to 11 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
cm
  Day 1 | 0.79 (1.54) | 0.00 (0.00)
  Days 1 to 11 | 0.51 (0.79) | 0.05 (0.17)
  Days 2 to 11 | 0.48 (0.82) | 0.05 (0.18)
  Day 2 | 0.46 (1.55) | 0.08 (0.48)
  Day 3 | 0.56 (1.47) | 0.03 (0.16)
  Day 4 | 0.41 (1.19) | 0.13 (0.47)
  Day 5 | 0.33 (1.11) | 0.00 (0.00)
  Day 6 | 0.56 (1.25) | 0.00 (0.00)
  Day 7 | 0.49 (1.47) | 0.03 (0.16)
  Day 8 | 0.67 (1.49) | 0.08 (0.35)
  Day 9 | 0.44 (1.23) | 0.10 (0.50)
  Day 10 | 0.59 (1.62) | 0.08 (0.35)
  Day 11 | 0.28 (1.45) | 0.03 (0.16)

22. Secondary Outcome: Change From Baseline in Body Weight
Description: The change in body weight collected at Day 12 relative to Baseline. A negative change from Baseline indicates a reduction in body weight and a positive change from Baseline indicates an increase in body weight.
Time Frame: Baseline and Day 12 of each period
Population: All participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
kilograms | 0.4 (0.95) | 0.1 (1.1)

23. Secondary Outcome: Change From Baseline in Hemoglobin
Description: The change in the value of hemoglobin collected at Day 12 relative to Baseline. A negative change from Baseline indicates a reduction in hemoglobin and a positive change from Baseline indicates an increase in hemoglobin.
Time Frame: Baseline and Day 12 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: grams/deciliter (mg/dL)
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
grams/deciliter (mg/dL) | -0.16 (0.68) | 0.14 (0.68)

24. Secondary Outcome: Number of Participants With Skin Rash
Time Frame: 11 days of each period
Population: All randomized participants who completed both periods of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
Participants | 0 | 0

25. Other Pre Specified Outcome: Reliability Index, Calculated as Percent of Possible Values Actually Recorded by CGM
Time Frame: 11 days
Population: All randomized participants who completed both periods.
Measure: Mean (Standard Deviation); unit: percentage of possible values
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
percentage of possible values | 96.6 (1.4) | 96.3 (1.6)

26. Other Pre Specified Outcome: Number of Unscheduled Infusion Set Replacements
Time Frame: 11 days
Population: All randomized participants who completed both periods of the study. Glucagon infusion sets are not applicable to the Usual Care arm.
Measure: Number; unit: Infusion Set Relacements
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
Infusion Set Relacements
  Glucagon Unscheduled Infusion Set Replacements: number analyzed (Participants) | 39 | 0
  Glucagon Unscheduled Infusion Set Replacements | 14 |
  Insulin Unscheduled Infusion Set Replacements | 11 | 15

27. Other Pre Specified Outcome: Mean Daily Basal Insulin Dose
Description: Daily basal insulin dose reported in Units per kilogram per day (U/kg/day).
Time Frame: Day 1, Days 2 to 11, each individual day 2 to 11 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
U/kg/day
  Day 1 | 0.3 (0.1) | 0.3 (0.1)
  Days 2 to 11 | 0.3 (0.1) | 0.3 (0.002)
  Day 2 | 0.3 (0.1) | 0.3 (0.1)
  Day 3 | 0.3 (0.1) | 0.3 (0.1)
  Day 4 | 0.3 (0.1) | 0.3 (0.1)
  Day 5 | 0.3 (0.1) | 0.3 (0.1)
  Day 6 | 0.3 (0.1) | 0.3 (0.1)
  Day 7 | 0.3 (0.1) | 0.3 (0.1)
  Day 8 | 0.3 (0.1) | 0.3 (0.1)
  Day 9 | 0.3 (0.1) | 0.3 (0.1)
  Day 10 | 0.3 (0.1) | 0.3 (0.1)
  Day 11 | 0.3 (0.1) | 0.3 (0.1)

28. Other Pre Specified Outcome: Mean Daily Bolus Insulin Dose
Description: Daily bolus insulin dose reported in Units per kilogram per day (U/kg/day).
Time Frame: Day 1, Days 1 to 11, Days 2 to 11, each individual day 2 to 11 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
U/kg/day
  Day 1 | 0.4 (0.1) | 0.3 (0.2)
  Days 1 to 11 | 0.4 (0.1) | 0.3 (0.015)
  Days 2 to 11 | 0.4 (0.1) | 0.3 (0.015)
  Day 2 | 0.4 (0.1) | 0.3 (0.2)
  Day 3 | 0.4 (0.1) | 0.3 (0.2)
  Day 4 | 0.4 (0.1) | 0.3 (0.3)
  Day 5 | 0.4 (0.1) | 0.3 (0.2)
  Day 6 | 0.4 (0.1) | 0.3 (0.2)
  Day 7 | 0.4 (0.1) | 0.3 (0.2)
  Day 8 | 0.4 (0.1) | 0.3 (0.2)
  Day 9 | 0.4 (0.1) | 0.3 (0.2)
  Day 10 | 0.4 (0.2) | 0.3 (0.2)
  Day 11 | 0.4 (0.1) | 0.3 (0.2)

29. Other Pre Specified Outcome: CGM Mean Absolute Relative Differences (MARD) Versus Time-stamped Blood Glucose (BG) Values From Meter Downloads
Description: This outcome measure compares the time stamped PG values from the glucose meter to the corresponding CGM glucose value to determine the overall accuracy of the CGM.
Time Frame: 11 days
Population: All randomized participants who completed both periods.
Measure: Mean (Standard Deviation); unit: percent difference
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 39 | 39
percent difference | 19.2 (31.4) | 18.0 (28.2)

ADVERSE EVENTS:
Time Frame: Days 1 to 11
Arm/Group | Bionic Pancreas | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 41/41 | 41/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bionic Pancreas (N=41) | Usual Care (N=41)
Hypoglycemia (Metabolism and nutrition disorders) | 41 | 41
Nausea (Gastrointestinal disorders) | 21 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No